CLINICAL TRIAL: NCT03792802
Title: EFFECT OF USING SAME DERMATOME LİNE FOR ALL PORT SİTES IN LAPAROSCOPIC APPENDECTOMY IN ACUTE APANDICITIS
Acronym: DERMATOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, asistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ANIL ERGIN..
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Appendicitis
Keywords: dermatome; laparoscopic appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: Model 1: Single dermatome laparoscopic appendectomy Model 2: Standard laparoscopic appendectomy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Care provider, participant and investigator did not know which type of surgery has applicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic port sites (Active Comparator): . Port sites located 1 infraumbilical , 1 right lower quadrant and 1 left lower quadrent
  Interventions: Procedure: laparoscopic appendectomy port sites
- same dermatome port sites (Active Comparator): One of the port will put in infraumbilical site and the other ones will put 10 cm right and left side from infraumbilical port.
  Interventions: Procedure: laparoscopic appendectomy port sites

INTERVENTIONS:
Procedure: laparoscopic appendectomy port sites — one group will have classic port sites ;.Port sites located 1 infraumbilical , 1 right lower quadrant and 1 left lower quadrent . one group will have same dermatome port sites ; One of the port will put in infraumbilical site and the other ones will put 10 cm right and left side from infraumbilical port
  Other Names: port sites in the same dermatome T10

SUMMARY:
Acute apandicitis is the one of most common cause of abdominal pain.Most of center still use open appendectomy(OA) technic for acute apandisitis.But Semm was defined Laparoskopic appendectomy(LA) with 3 ports in 1983.Today surgeons skill and experience ara increasing about LA day by day. Because of advantages of LA , this technical tend to be gold standart in acute apandisitis. In LA , all of centers use same technic as 3 ports for the surgery. Port sites located 1 infraumbilical , 1 right lower quadrant and 1 left lower quadrent in this surgery. But 3 dermatome lines have been effected in this style of location .This 3 points causes more pain postoperatively.In our study we will define the port locations into the same dermatome line (T10) . Purpose of this research is incerasing the postoperative pain score ,decreasing postoperative need of analgesia and develop the patient satisfy.

DETAILED DESCRIPTION:
Most of surgeon use 3 port sites for the Laparoscopic appendectomy in acute apandisitis. One of them places to infraumbilical region.,The other ports place to 1 right lower quadrant and 1 left lower quadrent routinly. In this study we will define T10 dermatome lregion in 40 patients who are planing to Laparoscopic appendectomy because of acute apandisitis older than 18 years old , before the surgery . All of LA port sites will put in this region .One of the port will put in infraumbilical site and the other ones will put 10 cm right and left side from infraumbilical port. In control group classic LA port sites will be used in the surgery for 40 patients.These two groups will compare after the surgery by Visual Analog Scala (VAS) Postoperative pain quantity will save by using VAS. Measurements will save in 1 hour,2 hour , 6 hour ,12 hour and 24 hour. All patients will take the same pain relief medication peroperatively and postoperatively. If the pain score would be more than 3 in VAS , all patient will take additional analgesic doses.Patients and VAS researcher will not know the patients group .Study will do as double blind.

ELIGIBILITY:
Inclusion Criteria:

* The patients who will undergo to Laparoscopic Appendectomy for Acute Apandisitis older than 18 years old.

Exclusion Criteria:

* Perforated apandisitis
* Plastrone apndisitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
compare of same dermatome trochar sites and different dermatomes trokar sites methods for postoperative pain relief by VAS (Visual Analog Scala) | 24 hours
  pain scores of the participants will be followed at postoperative 1,2,4,6,12,24 hour (up to 24 hours).
  (VAS: from 0 to 10, 0 = no pain, 10 = the worst pain) The higher score idicates the worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No